CLINICAL TRIAL: NCT04836819
Title: Comparison of Lidocaine, Dexmedetomidine and Ketamine in Multimodal Analgesia Management Following Sleeve Gastrectomy Surgery: A Randomized Double-Blind Trial
Brief Title: Analgesia Management in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Yasemin Burcu Ustun, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SGPAM-DKL11
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate; Pain; Postoperative
Keywords: Dexmedetomidine; Ketamine; Lidocaine; Obesity; Morbid; Pain; Postoperative
MeSH Terms: conditions — Obesity, Morbid; Pain; Obesity | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The patients will be randomly classified into three groups.
Who Masked: Participant, Investigator
Masking Description: Drugs to be used will be prepared 30 minutes before the surgery in the drug preparation room by a nurse who is not involved in the study. Investigators and patients will be blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group L (Active Comparator): IV lidocaine infusion (1-2 mg/kg/h) up to postoperative 12 hours.
  Interventions: Drug: Lidocain
- Group K (Active Comparator): IV ketamine infusion (0.3-0.5 mg/kg/h) up to postoperative 12 hours.
  Interventions: Drug: Ketamine
- Group D (Active Comparator): IV dexmedetomidine infusion (0.3-0.5 mg/kg/h) up to postoperative 12 hours.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Lidocain — IV lidocaine infusion (2 mg/kg/h) will be initiated after anesthesia induction and decrease the dosage to 1 mg/kg/h at the end of surgery. The infusion will continue until 12 hours after the operation.1 g paracetamol, 100 mg tramadol, 100 mg ketoprofen, and 4 mg dexamethasone will be administered to all patients pre-emptively. Granisetron (3 mg) will be administered 30 minutes before the end of surgery. In the postoperative period, i.v. Paracetamol will be administered at 8-hour intervals and 25-50 mg meperidine i.m. (maximum dose 200 mg) as rescue analgesia when requested by the patient and if VAS>4.
  Arms: Group L
Drug: Ketamine — IV ketamine infusion (0.5 mg/kg/h) will be initiated after anesthesia induction and decrease the dosage to 0.3 mg/kg/h at the end of surgery. The infusion will continue until 12 hours after the operation.1 g paracetamol, 100 mg tramadol, 100 mg ketoprofen, and 4 mg dexamethasone will be administered to all patients pre-emptively. Granisetron (3 mg) will be administered 30 minutes before the end of surgery. In the postoperative period, i.v. Paracetamol will be administered at 8-hour intervals and 25-50 mg meperidine i.m. (maximum dose 200 mg) as rescue analgesia when requested by the patient and if VAS>4.
  Arms: Group K
Drug: Dexmedetomidine — IV dexmedetomidine infusion (0.5 mg/kg/h) will be initiated after anesthesia induction and decrease the dosage to 0.3 mg/kg/h at the end of surgery. The infusion will continue until 12 hours after the operation.1 g paracetamol, 100 mg tramadol, 100 mg ketoprofen, and 4 mg dexamethasone will be administered to all patients pre-emptively. Granisetron (3 mg) will be administered 30 minutes before the end of surgery. In the postoperative period, i.v. Paracetamol will be administered at 8-hour intervals and 25-50 mg meperidine i.m. (maximum dose 200 mg) as rescue analgesia when requested by the patient and if VAS>4.
  Arms: Group D

SUMMARY:
Following laparoscopic bariatric surgery, multimodal analgesia is recommended to avoid the adverse effects of opioids by reducing their use. Although lidocaine, ketamine, and dexmedetomidine have been used as adjuvant analgesics, no studies have evaluated the superiority of their intra- and postoperative infusions as components of multimodal analgesia in bariatric surgery. The present study is aimed to compare lidocaine, dexmedetomidine, and ketamine in multimodal analgesia management following Sleeve Gastrectomy Surgery. Postoperative pain scores, the requirement for additional postoperative analgesia, retching, nausea and vomiting, time to mobilization, and hospital length of stay will be evaluated.

DETAILED DESCRIPTION:
Patients will be divided into three groups.

Group L: The patients will receive intravenous lidocaine (2 mg/kg/h) immediately after anesthesia induction. At the end of the surgery, the dose will be decreased to 1 mg/kg/h. The infusion will continue until 12 hours after the operation.

Group K: The patients will receive intravenous ketamine (0.5 mg/kg/h) immediately after anesthesia induction. At the end of the surgery, the dose will be decreased to 0.3 mg/kg/h. The infusion will continue until 12 hours after the operation.

Group D: The patients will receive intravenous dexmedetomidine (0.5 mg/kg/h) immediately after anesthesia induction. At the end of the surgery, the dose will be decreased to 0.3 mg/kg/h. The infusion will continue until 12 hours after the operation.

Ketamine, lidocaine, and dexmedetomidine doses will be calculated according to ideal body weight, lean body weight, and actual body weight, respectively.

Randomization will be performed using a computer-generated random number list, and a statement indicating the patient's group will be placed in a closed envelope numbered according to the result. Each patient will be asked to choose an envelope, and the patients will be assigned to the study according to the group mentioned in the envelope.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index>35 kg/m2
* The American Society of Anaesthesiologists (ASA) physical status class II III
* Patients who will undergo an elective laparoscopic sleeve gastrectomy (LSG)

Exclusion Criteria:

* refusal to participate
* allergy to the study drugs
* chronic kidney disease (creatinine>150 μmol/L)
* mental illness
* liver, respiratory or oncological disease,
* cardiac dysfunction (ejection fraction <40%),
* uncontrolled hypertension,
* preoperative analgesic use,
* chronic pain,
* history of alcohol or drug addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain: VAS scores at rest and movement | Up to 15 days after the surgery.
  Pain status at rest and movement will be assessed by VAS scores. The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (worst pain imaginable).

SECONDARY OUTCOMES:
Postoperative Rescue Analgesic Requirement | Up to three days after surgery
  After the end of surgery 25-50 mg meperidine (maximum dose 200 mg) will be administered i.m. as rescue analgesia when requested by the patient and if VAS>4. the Rescue analgesic dosage will be recorded.
Postoperative nausea, retching and vomiting | Up to 3 days after surgery.
  The number of patients who has complained of nausea, retching and vomiting will be recorded.
Time to first mobilization | Up to 24 hours after surgery.
  The patients first mobilization time after the operation will be recorded.
Time to discharge | Trough hospital stay, an average of 1 week.
  The length of hospital stay will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Koksal, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belcaid I, Eipe N. Perioperative Pain Management in Morbid Obesity. Drugs. 2019 Jul;79(11):1163-1175. doi: 10.1007/s40265-019-01156-3. PMID 31256367
- [Background] Feld JM, Hoffman WE, Stechert MM, Hoffman IW, Ananda RC. Fentanyl or dexmedetomidine combined with desflurane for bariatric surgery. J Clin Anesth. 2006 Feb;18(1):24-8. doi: 10.1016/j.jclinane.2005.05.009. PMID 16517328
- [Background] Laskowski K, Stirling A, McKay WP, Lim HJ. A systematic review of intravenous ketamine for postoperative analgesia. Can J Anaesth. 2011 Oct;58(10):911-23. doi: 10.1007/s12630-011-9560-0. Epub 2011 Jul 20. PMID 21773855
- [Background] Ciftci B, Ekinci M, Celik EC, Kaciroglu A, Karakaya MA, Demiraran Y, Ozdenkaya Y. Comparison of Intravenous Ibuprofen and Paracetamol for Postoperative Pain Management after Laparoscopic Sleeve Gastrectomy. A Randomized Controlled Study. Obes Surg. 2019 Mar;29(3):765-770. doi: 10.1007/s11695-018-3613-1. PMID 30474791
- [Background] Bamgbade OA, Oluwole O, Khaw RR. Perioperative Analgesia for Fast-Track Laparoscopic Bariatric Surgery. Obes Surg. 2017 Jul;27(7):1828-1834. doi: 10.1007/s11695-017-2562-4. PMID 28120147